CLINICAL TRIAL: NCT00580073
Title: A Phase II Trial of Neoadjuvant FOLFOX4 and Cetuximab for Localized Adenocarcinoma of the Rectum
Brief Title: Phase II Trial of Neoadjuvant FOLFOX4 and Cetuximab for Localized Adenocarcinoma of Rectum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO06207; NCI-2011-00476 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison); H-2007-0197 (Other: Institutional Review Board)
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2017-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): FOLFOX4 + Cetuximab
  Interventions: Drug: FOLFOX4; Drug: Cetuximab

INTERVENTIONS:
Drug: FOLFOX4 — oxaliplatin (85mg/m2 on days 1 and 15 of each cycle)+ 5FU Bolus (400mg/m2 on days 1, 2, 15, and 16 of each cycle) + 5FU CI (600mg/m2 on days 1, 2, 15, and 16 of each cycle) + Leucovorin (200mg/m2 on days 1, 2, 15, and 16 of each cycle)
  Other Names: Oxaliplatin (Eloxatin), 5FU (5-Fluorouracil) and Leucovorin (Folinic Acid)
Drug: Cetuximab — Cetuximab 400mg/m2 on day 1 only, 250mg/mr on days 8, 15, and 22 of each cycle.
  Other Names: Cetuximab (C225, Erbitux)

SUMMARY:
This study involves the use of Oxaliplatin, 5-Fluorouracil (5-FU), Leucovorin and Cetuximab, which are all medicines approved by the Food and Drug Administration (FDA) and are commercially available. This treatment regimen will possibly be combined with radiation before and/or after surgery depending on your response to the treatment. Their use in this exact combination is considered experimental. The purpose of this study is to find out how effective this combination of chemotherapy is as treatment for rectal cancer that has not spread to other parts of the body. The side effects and survival experienced by subjects receiving these drugs will also be evaluated. This is a phase II research study.

DETAILED DESCRIPTION:
Primary Objective:

- Down-staging of the tumor

Secondary Objectives:

* Pathologic response rate
* Tumor marker response
* Incidence of sphincter sparing surgery
* Progression-free survival
* Overall Survival

ELIGIBILITY:
Inclusion Criteria:

* All patients must have newly diagnosed, histologically proven adenocarcinoma of the rectum. Locally advanced T3, T4 or any T with N1, N2, staged by trans-rectal ultrasound.
* All patients must have an abdominal/pelvis CT scan or MRI confirming no evidence of distant metastases.
* Patients must have an ECOG PS ≤ 2
* Patient has signed informed consent
* Lower Age Limit: 18 years
* Upper Age Limit: No upper age limit
* Laboratory parameters:

  * Hgb: > 9.0 g/dl
  * ANC >1500/ul
  * Platelet >100,000/ul
  * Creatinine < 2x ULN
  * Bilirubin < 2x ULN
  * ALT < 2x ULN

Exclusion Criteria:

* Administration of any prior systemic anticancer therapy for colorectal cancer (eg, chemotherapy, antibody therapy, immunotherapy, gene therapy, vaccine therapy, cytokine therapy, angiogenesis inhibitors).
* Previous intra-arterial cytotoxic chemotherapy given as treatment for colorectal cancer.
* Previous pelvic radiotherapy.
* Known allergy or intolerance to oxaliplatin, 5-FU, cetuximab or leucovorin.
* Pregnant or breast-feeding women: female patients must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. All at-risk female patients must have a negative serum pregnancy test within 7 days prior to registration.
* Active inflammatory bowel disease, significant bowel obstruction, or chronic diarrhea (grade 2).
* Myocardial infarction or stroke within the previous 6 months, or ongoing unstable angina, symptomatic congestive heart failure, or serious uncontrolled cardiac dysrhythmia.
* Known human immunodeficiency virus (HIV) positivity or acquired-immunodeficiency-syndrome (AIDS)-related illness.
* No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer for which the patient has been disease-free for 3 years.
* Known CNS metastases
* Preexisting neuropathy > Grade 2
* Prior therapy which specifically and directly targets the EGFR pathway
* Prior severe infusion reaction to a monoclonal antibody
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure and cardiomyopathy with decreased ejection fraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Huie, M.D., Study Chair — UW Paul P. Carbone Comprehensive Cancer Center
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 4/08 and 11/09 from a large cancer research institution.
Groups:
- FOLFOX4 + Cetuximab: FOLFOX4: oxaliplatin (85mg/m2 on days 1 and 15 of each cycle)+ 5FU (5-fluorouracil) Bolus (400mg/m2 on days 1, 2, 15, and 16 of each cycle) + 5FU CI (600mg/m2 on days 1, 2, 15, and 16 of each cycle) + Leucovorin (200mg/m2 on days 1, 2, 15, and 16 of each cycle)
  Cetuximab: Cetuximab 400mg/m2 on day 1 only, 250mg/mr on days 8, 15, and 22 of each cycle.
Period: Overall Study
Arm/Group | FOLFOX4 + Cetuximab
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FOLFOX4 + Cetuximab: FOLFOX4: oxaliplatin (85mg/m2 on days 1 and 15 of each cycle)+ 5FU Bolus (400mg/m2 on days 1, 2, 15, and 16 of each cycle) + 5FU CI (600mg/m2 on days 1, 2, 15, and 16 of each cycle) + Leucovorin (200mg/m2 on days 1, 2, 15, and 16 of each cycle)
  Cetuximab: Cetuximab 400mg/m2 on day 1 only, 250mg/mr on days 8, 15, and 22 of each cycle.
Arm/Group | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Down-staging of the Tumor; Response to Therapy
Description: Down-staging of the tumor and tumor response rate is defined as the proportion of participant who have any evidence of complete response (CR), pathologic complete response (pCR), or partial response (PR).
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 6
participants
  PR | 4
  pCR | 1
  CR | 0

2. Secondary Outcome: Progression Free Survival
Description: Number of participants who achieve progression free survival, defined as the time from date of registration to date of disease progression, up through study closure. Progressive disease is defined as ≥ 20% increase in the sum of the longest dimensions of the primary lesion taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 6
participants | 5

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of registration to date of death. In the absence of confirmation of death, survival time will be censored at the last date of follow-up.
Time Frame: Up to 3 years
Population: This study was closed because of withdrawal of funding. All participants were off study on 02/03/2011.
Arm/Group | FOLFOX4 + Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 of treatment through the Study Completion Date (02/03/2011), which is a time period of up to 3 years.
Description: Participants were closely monitored for treatment-related adverse events, especially infusion reactions, during the infusion and the post-infusion observation hour. All
Arm/Group | FOLFOX4 + Cetuximab
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX4 + Cetuximab (N=6)
Grade 3/4 neutropenia (Blood and lymphatic system disorders) | 3 (3)
Grade 3/4 potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Grade 3/4 neuropathy (Nervous system disorders) | 1 (1)
Grade 3/4 fatigue (General disorders) | 1 (1)
Grade 3/4 aspartate aminotransferase (AST) (Investigations) | 1 (1)
Grade 3/4 alanine aminotransferase (ALT) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX4 + Cetuximab (N=6)
Grade 1/2 rash (Skin and subcutaneous tissue disorders) | 4 (4)
Grade 1/2 neuropathy (Nervous system disorders) | 3 (3)
Grade 1/2 neutropenia (Blood and lymphatic system disorders) | 3 (3)
Grade 1/2 fatigue (General disorders) | 3 (3)
Grade 1/2 mucositis (Gastrointestinal disorders) | 2 (2)
Grade 1/2 nausea (Gastrointestinal disorders) | 2 (2)
Grade 1/2 diarrhea (Gastrointestinal disorders) | 2 (2)
Grade 1/2 potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Grade 1/2 aspartate aminotransferase (AST) (Investigations) | 1 (1)
Grade 1/2 alanine transaminase (ALT) (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed due to withdrawal of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes